CLINICAL TRIAL: NCT05756803
Title: Changes in Penile Firmness With Low-Intensity Shockwave Therapy (LiST)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-1144
Record Dates: First submitted 2021-10-19; First posted 2023-03-06 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Low Intensity Acoustic Shockwave Therapy (Experimental): The device applies a low-intensity shockwave to the surface of the penis using an ultrasound gel as the coupling agent. The low-intensity shockwave therapy device will be used with the purpose of improving penile blood flow and restoring sexual function in men with impaired erectile function.
  Interventions: Device: Low-intensity acoustic shockwave therapy

INTERVENTIONS:
Device: Low-intensity acoustic shockwave therapy — The study is being done to find out if low-intensity shockwave therapy can improve penile blood flow and restore sexual function in men with impaired erectile function.

SUMMARY:
Patients presenting with erectile dysfunction are often found to have increased corporal firmness on elastography. We hypothesize that this corporal firmness reflects reversable changes that can be altered by Low-Intensity Shockwave Therapy (LiST). In this pilot study patients found to have increased corporal firmness will be treated with LiST.

DETAILED DESCRIPTION:
This study will enroll men between the ages of 18 and 65 with corporal cavernosal firmness on elastography. The participants study duration is 3 months long and includes eight visits at the study center. Study visits consist of physical exam, vital signs, questionnaires, blood draws, and administration of low-intensity shockware therapy (LiST).

Low intensity extracorporeal (i.e., outside the body) shockwave therapy (LiST) is a treatment that has been in use since 2010 and has become commonly used Internationally and in the United States since 2015. The device applies a low-intensity shockwave to the surface of the penis using an ultrasound gel as the coupling agent.

The study will evaluate changes in corporal cavernosal firmness and changes in penile vascular blood flow.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Men aged 18-64
4. Sexually active men and evidence of increased firmness on elastography during their standard evaluation for erectile dysfunction.

Exclusion Criteria:

1. Within two weeks of Visit 1 using erectogenic medications including PDE5 inhibitors and/or penile injection therapy
2. Presence of a penile implant.
3. Presence of cardiac pacemaker or defibrillator
4. Patients who are using devices which are sensitive to electromagnetic radiation.
5. Screening ultrasound positive for testicular cancer
6. Presence of untreated prostate cancer
7. Patients with severe coagulation disorders
8. Patient that in the opinion of the Principal Investigator would be non-compliant with the study

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Men aged 18-64
Enrollment: 20 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate changes in corporal cavernosal firmness with Low-Intensity Acoustic Shockwave Therapy (LiST) | 12 Weeks
  Change in corporal firmness (KPa) with Low-Intensity Acoustic Shockwave Therapy (LiST)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Private Office, Great Neck, New York
  - The Smith Institute for Urology, Lake Success, New York